CLINICAL TRIAL: NCT03453645
Title: Modification of Rhythmic Risk Assessment by Ventricular Tachycardia Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0066; 2017-A00582-51 (Other: ID-RCB)
Record Dates: First submitted 2017-07-27; First posted 2018-03-05 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Ventricular Tachycardia
Keywords: ablation; sudden death; signal averaged ECG; T wave alternans; heart rate variability
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ventricular tachycardia ablation — The usual organization of hospitalization of the patients addressed for ventricular tachycardia ablation and his follow-up are not modified by the protocol. .

SUMMARY:
Sudden cardiac death is a frequent cause of cardiovascular mortality. Numerous rhythmic risk assessment criterion have been described targeting the substratum, the cardiac nervous tone or the trigger of arrhythmias. Development of ventricular tachycardia ablation in the past few years show interesting results preventing the recurrence of ventricular arrhythmias.

DETAILED DESCRIPTION:
Sudden cardiac death is a frequent cause of cardiovascular mortality. Numerous rhythmic risk assessment criterion have been described targeting the substratum, the cardiac nervous tone or the trigger of arrhythmias. Development of ventricular tachycardia ablation in the past few years show interesting results preventing the recurrence of ventricular arrhythmias.

Rhythmic risk assessment criterions have never been studied in relation with ventricular tachycardia ablation. The purpose of this study is to explore the modifications of these criterions after ventricular tachycardia ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ventricular tachycardia,
* patients with ischemic cardiomyopathy according to European Society of Cardiology Guidelines,
* patients with implanted cardiac defibrillator.

Exclusion Criteria:

* Contra-indication to stress test,
* permanent atrial fibrillation,
* permanent ventricular pacing,
* left bundle block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people wich an Ventricular Tachycardia Ablation necessary and programed
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
measure assessing change before and after Ventricular Tachycardia Ablation of the non-invasive parameters analysis of the rhythmic risk before and after Ventricular Tachycardia Ablation | 10 minutes and 60 minutes after the Ventricular Tachycardia Ablation
  non invasive parameters analysis of the rhythmic risk will be evaluated by the evaluation of the T wave alternans

SECONDARY OUTCOMES:
Assessing the correlations of the modifications of the risk criterion after ablation with the recurrences of arrhythmias at one year follow-up | 3 months, 6 months and 12 months after the Ventricular Tachycardia Ablation
  the recurrences of arrhythmias will be evaluated . There will be assessed by the informations reveled by the Implantable automatic defibrillator
Study of the correlation between the modifications of non-invasive parameters analysis of the rhythmic risk and the success of the ablation procedure | 3 months, 6 months and 12 months after the Ventricular Tachycardia Ablation
  Success of the ablation procedure is defined by the absence of inducible Ventricular Tachycardia at the end of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAURY, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France